CLINICAL TRIAL: NCT04292353
Title: Cerebral Morbidity After Radiation Therapy for Brain Tumors
Acronym: WP-12
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Morten Høyer, Professor, University of Aarhus
Other Study IDs: WP-12
Record Dates: First submitted 2018-06-01; First posted 2020-03-03 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Brain Tumor; Cognitive Impairment; Radiation Toxicity
Keywords: Brain tumor; Cognitive function; Radiation Therapy; Hippocampus
MeSH Terms: conditions — Brain Neoplasms; Cognitive Dysfunction; Radiation Injuries | interventions — Neuropsychological Tests; Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cognitive tests and Patient Reported Outcome

SUMMARY:
This study will assess cognitive function in patients with a primary brain tumour treated with radiation therapy (RT) to generate radio-sensitivity and volume effect parameters for the development of cognitive dysfunction. All types of brain tumours apart from glioblastoma will be included.

DETAILED DESCRIPTION:
RT to brain tumours causes cognitive dysfunction. The extent of RT induced changes in cognitive function and radio-sensitivity of the brain is unknown. RT with protons instead of photons spares the healthy brain tissue more and is believed to reduce the risk of cognitive dysfunction. There is modest knowledge on which parts of the brain we need to spare, to prevent cognitive dysfunction.

The study is a prospective nationwide study including approximately 60 brain tumour patients from the four neuro oncology centres in Denmark. The patients will do patient reported outcome (PRO) and undergo neuropsychological assessment with standardized tests: They will do this prior to RT treatment and ½, 1, 3 and 5 years afterwards. The PRO's included measures on quality of life, fatigue, sleep, depression, anxiety, and socio demografica. The standardized tests are: Trail making Test (TMT); Hopkins Verbal Learning Test (HVLT); Controlled Oral Word Association Test (COWAT) - Animals and S; Coding and Digit Span from WAIS-IV; Paced Auditory Serial Addition Test (PASAT). The correlation between cognitive scores and RT dose-volume parameters to specific areas in the brain will be tested.

This study will elucidate the dose-response relationship in radiation-induced damage to substructures of the brain such as hippocampus, thalamus, temporal and frontal lobes that will allow the clinician to prioritize these structures in planning of proton radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older and Danish speaking.
* Performance status WHO 0-2
* Capable of cooperating on testing
* Tumor histology (WHO 2016 classification) of the following types: anaplastic astrocytoma (IDH mutant), diffuse astrocytoma (IDH-mutant), gemistocytic astrocytoma (IDH mutant), diffuse astrocytoma (NOS), oligidendroglioma, meningioma, medulloblastoma (NOS), pituitary adenoma, other brain tumours including skull base sarcomas

Exclusion Criteria:

* Glioblastoma
* Performance status 3-4

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients will be diagnosed with a primary brain tumour and referred to radiation therapy. They will be recruited from the four neuro oncology centers in Denmark
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Impairment of memory as assessed by the HVLT-r test | 5 Years
  Examined by the Hopkins Verbal Learning Test. It will be correlated to the mean radiation dose to the hippocampus. Outcome is number of correct words (0-24)

SECONDARY OUTCOMES:
Processing speed | 5 Years
  Examined by the Trail making Test part A (TMT_A) and the Coding from WAIS-IV. Outcome for TMT_A is time in seconds (0-120 seconds). Outcome for Coding is number of correct (within 2 minutes) (0-100)
Attention and working memory | 5 Years
  Examined by WAIS_IV_digit_span and PASAT (Pased Auditory Seriel Addition Test). Outcome on WAIS digit span is number of correct (0-36) and outcome for PASAT is number of incorrects (0-60)
Verbal learning and memory | 5 Years
  Examine by the Hopkins Verbal Learning Test (HVLT) - total and delayed. Outcome is number of correct words (0-24)
Verbal fluency | 5 Years
  Examined by the Controlled Oral Word Association Test (COWAT) - Animals and letter_S. Outcome is number of words produced in 1 minute (0-100)
Executive function | 5 Years
  Examined by Trail making Test part B (TMT-B) and the STROOP colour and word test (STROOP). Outcome for TMT_B is time in seconds (0-300). Outcome for STROOP is number of corrects (0-120)
Global Health - Quality of life | 5 Years
  Assessed by questionnaire; EORTC QlQ-C30 in order to examine the level of quality of life in brain tumour patients who has received radiation therapy. Quality of life will be assessed by EORTC QIQ-C-30
Fatigue | 5 years
  Assessed by questionnaire: FACIT-Fatigue scale (version 4) in order to explore the level of fatigue in brain tumour patients who has received radiation therapy.
Qulity of Sleep | 5 years
  Assessed by questionnaire:Pittsburg Sleep Quality INDEX, PSQI in order to explore the level of quality of sleep in brain tumour patients who has received radiation therapy
Depression/Anxiety | 5 years
  Assessed by questionnaire: Hospital anxiety and depression Scale (HADS) in order to explore level of depression and anxiety in patients treated with radiation therapy for their brain tumour
Patient's Assessment of Own Functioning Inventory | 5 years
  Assessed by questionnaire; Patient's Assessment of Own Functioning Inventory (PAOFI), in order to assess patients own perception of cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Morten Høyer, M.D, Principal Investigator — Danish Center for Particel Therapy, Aarhus University Hospital, Denmark
Locations (4):
- Denmark (4):
  - Rigshospital, Copenhagen, Region H
  - Department of Oncology, Aarhus, Region Midt
  - Aalborg University Hospital, Aalborg, Region Nord
  - Odense University Hospital, Odense, Region Syd

IPD SHARING:
Plan to Share IPD: No